CLINICAL TRIAL: NCT01932294
Title: Medical Arm of the Interagency Registry for Mechanically Assisted Circulatory Support
Acronym: Medamacs
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Medamacs
Record Dates: First submitted 2013-04-12; First posted 2013-08-30 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2017-01

CONDITIONS: Heart Failure; Systolic Heart Failure
Keywords: Advanced Heart Failure; Refractory Heart Failure; Mechanical Circulatory Support Device; Ventricular Assist Device; Medamacs
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MedaMACS participants: All participants who have met the inclusion criteria.

SUMMARY:
Medamacs is a prospective, observational study of ambulatory patients with advanced heart failure. The study enrolls patients who have not yet received a Left Ventricular Assist Device (LVAD) but who receive their care at a hospital with a Joint Commission certified mechanical circulatory support program.

Medamacs is funded through the Interagency for Mechanically Assisted Circulatory Support (INTERMACS) NHLBI Contract.

DETAILED DESCRIPTION:
Participants between 18 and 80 years old with low ejection fraction history and hospitalization for heart failure within the past year will be screened for the study. All subjects who have been admitted to the heart failure service will be screened and recruited, either as an inpatient or during their first outpatient follow-up appointment by the investigator and research staff caring for patients in the advanced heart failure program.

Eligibility for enrollment will be based only upon information that is clinically available at the time of screening. The history of prior hospitalizations will be available from clinical records.

Routine evaluation and triage of ambulatory patients with advanced heart disease includes echocardiography and functional assessment with peak oxygen consumption and frequently 6 minute walk distance. The elements of information required for estimation of the Seattle Heart Failure Risk score will be gleaned from laboratory data, or imputed as described in the Seattle score literature. The research coordinator will enter this data onto a currently available website for calculation of the Seattle score.

Eligibility will be determined by the inclusion and exclusion criteria and the study research team will approach individual subjects who are potential candidates for participation once the subject's primary physician has given permission to approach. Only persons with a scientific or ethical reason will be excluded. Incarcerated prisoners have been excluded by this protocol.

Participants will be followed every 6 months for 24 months after two baseline visits. The 6 month and 18 month follow ups consist of telephone interviews. Follow ups at 12 months and 24 months consists of routine clinical visits.

Approximately 350 patients from 12 centers in the United States will be enrolled over a 12 month period.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with Advanced Heart Failure

1. Age 18-80 years
2. New York Heart Association class III-IV heart failure for 45 of the last 60 days
3. Left ventricular ejection fraction ≤ 35%
4. Heart failure diagnosis or typical symptoms for 12 months
5. Use of evidence based oral medications (beta-blockers, ACE-inhibitors/ARBs, aldosterone antagonist) for at least 3 months prior to enrollment or documented medication contraindication or intolerance.
6. Hospitalization for heart failure within the previous 12 months (other than for elective procedure)
7. Informed consent given

In Addition, they must have at least one of the following:

An additional unplanned hospitalization during the previous 12 months for a total of at least 2 inpatient hospitalizations lasting >24 hours with heart failure as the primary or secondary diagnosis within the previous 12 months

OR

1. Peak oxygen uptake (VO2) <55% of age- and sex-predicted (using Wasserman equation) OR a peak VO2 ≤16 ml/kg/min for men and ≤14 ml/kg/min for women in a test with an RER >1.08 on cardiopulmonary exercise testing.
2. 6-minute walk distance <300 meters without non-cardiac limitation.
3. Serum BNP > 1000 (NT-proBNP > 4000 pg/ml) as outpatient or at hospital discharge.

OR

Seattle Heart Failure Model Score > 1.5.

EXCLUSION CRITERIA:

1. Age >80 years or <18 years
2. Non-cardiac diagnosis anticipated to limit 2-year survival (≥30-50% mortality within 2 years from non-cardiac diagnosis)
3. Primary functional limitation from non-cardiac diagnosis even if not likely to limit survival
4. QRS > 120msec and planned biventricular pacemaker implant or biventricular pacemaker implantation within past 90 days
5. Current home intravenous inotrope therapy
6. Chronic hemodialysis or peritoneal dialysis
7. Scheduled for non-ventricular assist device cardiac surgery on current hospital admission
8. Obvious anatomical or other major contra-indication to any cardiac surgery in the future (e.g. previous pneumonectomy, advanced connective tissue disease)
9. Actively listed for heart transplant as UNOS Status 1 or 2
10. History of cardiac amyloidosis
11. Dominant lesion of at least moderate aortic or mitral stenosis or congenital structural heart defect.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be screened for this study if they are between 18 and 80 years old with low ejection fraction history and hospitalization for heart failure within the past year. All subjects who have been admitted to the heart failure service will be screened and recruited for study participation, either as an inpatient or during their first outpatient follow-up appointment by the investigator and research staff caring for patients in the advanced heart failure program of the enrolling center.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Kirklin, MD, Principal Investigator — INTERMACS Principal Investigator
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Beverly Hills, California
  - University of Colorado, Aurora, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) is not available. De-identified datasets may be available upon approval.

REFERENCES:
- [Background] Kirklin JK, Naftel DC, Kormos RL, Stevenson LW, Pagani FD, Miller MA, Baldwin JT, Young JB. Fifth INTERMACS annual report: risk factor analysis from more than 6,000 mechanical circulatory support patients. J Heart Lung Transplant. 2013 Feb;32(2):141-56. doi: 10.1016/j.healun.2012.12.004. PMID 23352390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MedaMACS Participants
Started | 171
Completed | 72
Not Completed | 99
Not completed — Death | 43
Not completed — Lost to Follow-up | 8
Not completed — VAD Implantation | 20
Not completed — Heart Transplantation | 16
Not completed — Transferred to other hospitals | 12

BASELINE CHARACTERISTICS:
Arm/Group | MedaMACS Participants
Number analyzed (Participants) | 171
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant missed this variable
  Participants
    number analyzed (Participants) | 170
    <=18 years | 0
    Between 18 and 65 years | 53
    >=65 years | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.03 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant missing a value for the variable
  Participants
    number analyzed (Participants) | 170
    Female | 57
    Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 160
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 119
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 171

OUTCOME MEASURES:

1. Primary Outcome: Number of Heart Failure Participants Deceased at 24 Months
Description: Death after the baseline visit up to 24 months
Time Frame: 6 month intervals after the baseline visit up to 24 months
Population: By the end of the follow-up, 43 patients had deceased.
Measure: Count of Participants; unit: Participants
Groups:
- MedaMACS Participants: All participants who have met the inclusion criteria. By the end of the follow-up, 43 out of 171 patients died.
Arm/Group | MedaMACS Participants
Number analyzed (Participants) | 171
Participants | 43

2. Secondary Outcome: Number of Participants With Known Ventricular Assist Device (VAD) Implantation
Description: Known VAD implantation after the baseline visit up to 24 months
Time Frame: 6 month intervals after the baseline visit up to 24 months
Population: Patients with known endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | MedaMACS Participants
Number analyzed (Participants) | 171
Participants | 20

3. Secondary Outcome: Number of Participants With Known Heart Transplantation
Description: Heart transplantation after the baseline visit up to 24 months
Time Frame: 6 month intervals after the baseline visit up to 24 months
Population: Patients with known endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | MedaMACS Participants
Number analyzed (Participants) | 171
Participants | 16

ADVERSE EVENTS:
Time Frame: After the baseline visit and up to 24 months
Arm/Group | MedaMACS Participants
All-Cause Mortality (participants affected / at risk) | 43/171
Serious Adverse Events (participants affected / at risk) | 93/171
Other Adverse Events (participants affected / at risk) | 12/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedaMACS Participants (N=171)
Rehospitalization (Investigations) | 93 (273) — All-cause Rehospitalizations
IV Inotropes Dependent at 6 months (Cardiac disorders) | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedaMACS Participants (N=171)
All-location Infection (Infections and infestations) | 12 (19) — All-location Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT01932294/Prot_SAP_000.pdf